CLINICAL TRIAL: NCT01514526
Title: Phase II Clinical Trial of Dovitinib (TKI-258) in First-line Metastatic or Locally Advanced Non-resectable Adrenocortical Carcinoma
Brief Title: Clinical Trial of Dovitinib in First-line Metastatic or Locally Advanced Non-resectable Adrenocortical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG2011-03; 2011-002873-47 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2012-01-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-04

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib (Experimental): Dovitinib (TKI-258) f 500 mg / day (5 x 100mg) once daily. The patient will continue on treatment until disease progression,unacceptable toxicity, death or premature withdrawal.
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Dovitinib (TKI-258), gelatin capsule of 100mg, developed and supplied by Novartis Inc. The study regimen consists of the administration of 500 mg / day (5 x 100mg) once daily, taken orally with a large amount of water, preferably one hour prior to a meal or at least two hours following a meal. This dose will be taken once daily according to 5 days on/2 days off schedule.
  The patient will continue on treatment until disease progression,unacceptable toxicity, death or premature withdrawal.
  Other Names: TKI258

SUMMARY:
* Design: non-randomized, open label, phase II clinical trial.
* Study population and disease: adult patients with metastatic or locally advanced non-resectable adrenocortical carcinoma, confirmed histologically.
* Estimated number of patients: 15.
* Study drug: dovitinib (TKI-258), dosed on a flat scale of 500mg/day on a 5 days on / 2 days off.
* Treatment duration: study treatment period will be continued until disease progression, unacceptable toxicity, death or premature withdrawal from study. An average of 6 months treatment period is expected.
* Study duration: expected recruitment period will be 18 months, and patients will be followed for 6 additional months after last patient is included in the trial.Study total expected duration is 24 months.
* Sites: the study is planned to be conducted in 7 Spanish centers.

DETAILED DESCRIPTION:
Non applicable

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* A performance status of 0, 1, or 2, according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Histologically confirmed adrenocortical carcinoma.
* Metastatic or locally advanced non-resectable disease.
* At least one radiologically measurable lesion, according to RECIST 1.1.
* Adequate liver function as shown by: serum or plasma ALT and AST ≤ 3.0 x ULN (regardless of the presence or absence of metastases)and serum or plasma total bilirubin: ≤ 1.5 x ULN.
* Adequate bone marrow function as shown by: blood absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L and hemoglobin (Hb) > 9g/dL.
* Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN.
* Patients give a written informed consent obtained according to local guidelines.

Exclusion Criteria:

* Prior chemotherapy other than mitotane (Patients who have previously received mitotane will only be eligible if drig has been withdrawn at least two weeks earlier than dovitinib first dose is administered).
* Patients with another primary malignancy within 3 years prior to starting the study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or completely excised basal or squamous cell carcinoma of the skin.
* Patients who have received radical radiotherapy ≤4 weeks prior to starting the study treatment or who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤2 weeks prior to starting study treatment is allowed.
* Patients who have undergone any major surgery (i.e., intra-thoracic, intrabdominal, or intra-pelvic) ≤4 weeks prior to starting study treatment or who have not recovered from side effects of such therapy.
* Patients with a history of pulmonary embolism (PE) within the past 6 months or untreated deep-venous-thrombosis (DVT) within the past 6 months. Adequately treated DVT will be permitted providing that patient has been on anticoagulation for at least 2 weeks.
* Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias.
  * Clinically significant resting bradycardia.
  * LVEF <45% when assessed by 2-D echocardiogram (ECHO) or multiple gated acquisition scan (MUGA). (No basal cardiac test is mandatory other than ECG)
  * Any of the following within 6 months prior to starting study treatment: Myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF),Cerebrovascular Accident (CVA), Transient Ischemic Attack TIA).
  * Uncontrolled hypertension defined by a SBP ≥160 mm Hg and/or DBP ≥100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication (s) is allowed prior to study entry.
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Dovitinib (TKI258) (i.e., severe ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive (>1m) small bowel resection, inability to swallow oral medications). Prior partial or total gastrectomy is not an exclusion criterion.
* Known diagnosis of human immunodeficiency virus (HIV) infection. HIV testing is not mandatory.
* Patients who are currently receiving full dose of anticoagulation treatment with therapeutic doses of dicumarinical drugs as warfarin/acenocoumarol or anti-platelet therapy (i.e.,clopidogrel bisulfate). Treatment with acetylsalicyclic acid 100mg daily is allowed, as well as prophylactic or therapeutic low-weight-heparin.
* Pregnant or breast-feeding women.
* Women of child-bearing potential not employing an effective method of birth control. Effective contraception (e.g. condom with spermicidal jelly, foam suppository or film; diaphragm with spermicide; male condom and diaphragm with spermicide) must be used throughout the trial and 8 weeks after the end of Dovitinib treatment. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study drug. Women of child-bearing potential not employing and not willing to use an effective method of birth control. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Fertile males not willing to use contraception as stated above.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Efficacy | Up to 6 months (Study treatment expected duration)
  Efficacy in terms of overall response rate (ORR) of dovitinib as treatment for metastatic or locally advanced non-resectable primary adrenocortical carcinoma (measured by an external evaluator)

SECONDARY OUTCOMES:
Safety profile of dovitinib in study population | Up to 24 months (Study expected duration, including patient treatment and follow up)
  Safety will be assessed considering the number of study participants with Adverse Events during the conduct of the trial, from date of patient inclusion until the date of study end, up to 24 months.
Efficacy of dovitinib in reducing ACC hormonal production (cortisol, testosterone, aldosterone or estrogens) | Up to 6 months (Study treatment expected duration)
  Efficacy of dovitinib in reducing ACC hormonal production (cortisol, testosterone, aldosterone or estrogens)
Progression free survival (PFS) in all treated patients (measured by an external evaluator) | Up to 24 months (Study expected duration, including patient treatment and follow up)
  From date of patient inclusion until the date of first documented progression, assessed up to 24 months.
Overall survival (OS)(measured by an external evaluator) | Up to 24 months (Study expected duration, including patient treatment and follow up)
  From date of patient inclusion until the date of of death from any cause, assessed up to 24 months.
Quality of Life (QoL) | Up to 24 months (Study expected duration, including patient treatment and follow up)
  From date of patient inclusion until the date of study end, up to 24 months.
Progression Free Survival and Overall Survival (determined by the local researchers) | Up to 24 months (Study expected duration, including patient treatment and follow up)
  From date of patient inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García-Donás Jiménez, MD, Principal Investigator — Spanish Oncology Genito-Urinary Group
Locations (7):
- Spain (7):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Fundación Instituto Valenciano de Oncología, Valencia

REFERENCES:
- See also: Spanish Oncology Genitourinary Group - Sponsor site — http://www.sogug.es